CLINICAL TRIAL: NCT02310958
Title: A Single Center, Retrospective Study of the Outcome of Laparoscopic Inguinal Herniorraphy in Children
Brief Title: Outcome of Laparoscopic Inguinal Herniorraphy in Children
Status: Completed | Type: Observational
Sponsor: Johannes Mayr (Other)
Responsible Party: Sponsor-Investigator, Johannes Mayr, Professor, University Children's Hospital Basel
Organization: University Children's Hospital Basel (Other)
Other Study IDs: EKNZ2014-247
Record Dates: First submitted 2014-11-30; First posted 2014-12-08 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Hernia, Inguinal
Keywords: Lapraroscopic surgical procedure; infant; complications; inguinal hernia; hernia recurrence
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with inguinal hernia: Laparoscopic surgical hernia repair in children aged between 1 day and 16 years
  Interventions: Procedure: Laparoscopic surgical hernia repair

INTERVENTIONS:
Procedure: Laparoscopic surgical hernia repair — Laparoscopic surgical hernia repair in children

SUMMARY:
The investigators plan a retrospective, single-center outcome analysis of laparoscopic hernia repair in children operated between March 2nd, 2010, and March 1st, 2014. Data analysis will be based on a review of hospital records and a questionnaire answered by families. Patient demographics (age, gender), affected side, type and duration of laparoscopic intervention, and outcome parameters (hernia recurrence, post-operative complications, eg. infections, length and type of postoperative pain medication, and length of the postoperative hospital stay) will be analysed.

DETAILED DESCRIPTION:
Hernias of the abdominal wall occur if intra-abdominal tissue or peritoneum bulges through the abdominal wall. The most frequent locations of abdominal wall hernia are the inguinal region close to the groin, the umbilicus, and scars. Congenital inguinal hernias occur more frequently in the inguinal region if the vaginal process is not closed adequately at birth. Surgical procedures for correction of inguinal hernias are frequently carried out in children. Laparoscopic procedures to correct inguinal hernias in children are gaining more acceptance. The laparoscopic closure of hernias in children is considered effective and safe and represents an accepted alternative to the open surgical hernia repair. When compared to open surgical hernia repair in children, laparoscopic hernia repair causes smaller scars, allows for a faster postoperative recovery of children, requires less pain medication, and allows for an inspection of the contralateral side, thus facilitating simultaneous hernia repair in the same operation.

We aim to investigate the short-term results of laparoscopic inguinal hernia repair in children. The main outcome parameter of this single-center study is hernia recurrence or the occurrence of contralateral metachronous hernia. Secondary outcome measures are postoperative complications such as infections of the wound regions, the time between operation and discharge from hospital, and postoperative pain medication requirements. We chose a 4-year time interval for inclusion of patients. Data are retrieved from hospital records in a retrospective evaluation. In addition, a structured questionnaire sent to the families of children will document postoperative complaints and complications from 3 months after the operation onwards. Families not responding to the questionnaire will be offered a structured telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 day and 16 years who underwent a laparoscopic surgical procedure for correction of unilateral or bilateral inguinal hernia or recurrent inguinal hernia at a single institution

Exclusion Criteria:

* age of patient more than 16 years
* patients suffering from neuromuscular, chronic abdominal, chronic pulmonary, or malignant disorders
* patients suffering from degenerative soft tissue disorders
* patients receiving immunosuppressive drugs for more than 3 weeks or during a - 3-week perioperative time interval

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 1 day and 16 years who underwent laparoscopic surgical inguinal hernia repair between March 2010 and March 2014 at a single institution.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Inguinal hernia recurrence | Participants will be followed for 3 months up to 51 months after the surgical procedure, an expected average of 27 months

SECONDARY OUTCOMES:
postoperative complications (infections) | Participants will be followed for 3 months up to 51 months after the surgical procedure, an expected average of 27 months
length of hospital stay | Participants will be followed for 3 months up to 51 months after the surgical procedure, an expected average of 27 months
type of pain medication and duration of use after surgical procedure | Participants will be followed for 3 months up to 51 months after the surgical procedure, an expected average of 27 months
metachronous hernia occurrence | Participants will be followed for 3 months up to 51 months after the surgical procedure, an expected average of 27 months
  Occurrence of contralateral hernia after operation of unilateral hernia

CONTACTS AND LOCATIONS:
Overall Officials: Sucharitha Geiger, Study Chair — University Childrens Hospital Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Surgeons. Surgical Patient Education. http://www.facs.org/patient education.
- [Background] Kapur P, Caty MG, Glick PL. Pediatric hernias and hydroceles. Pediatr Clin North Am. 1998 Aug;45(4):773-89. doi: 10.1016/s0031-3955(05)70044-4. PMID 9728185
- [Background] Kiesewetter WB, Oh KS. Unilateral inguinal hernias in children: What about the opposite side? Arch Surg. 1980 Dec;115(12):1443-5. doi: 10.1001/archsurg.1980.01380120019005. PMID 7447688
- [Background] Ramshaw BJ, Esartia P, Schwab J, Mason EM, Wilson RA, Duncan TD, Miller J, Lucas GW, Promes J. Comparison of laparoscopic and open ventral herniorrhaphy. Am Surg. 1999 Sep;65(9):827-31; discussion 831-2. PMID 10484084
- [Background] Tsai YC, Wu CC, Yang SS. Minilaparoscopic herniorrhaphy with hernia sac transection in children and young adults: a preliminary report. Surg Endosc. 2007 Sep;21(9):1623-5. doi: 10.1007/s00464-007-9207-y. Epub 2007 Mar 13. PMID 17353989
- [Background] Tsai YC, Wu CC, Yang SS. Is local anesthesia or oral analgesics necessary after mini-laparoscopic functional surgery in children and young adults?: A prospective randomized trial. Surg Laparosc Endosc Percutan Tech. 2008 Aug;18(4):344-7. doi: 10.1097/SLE.0b013e318172ab33. PMID 18716531